CLINICAL TRIAL: NCT04957654
Title: A Comparative Study Evaluating Vestibular Socket Therapy in Immediate Implants Using Different Grafting Materials
Brief Title: Vestibular Socket Therapy in Immediate Implants With Grafting Materials
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Mohamed Mofreh Hamada Hamed (Other)
Responsible Party: Sponsor-Investigator, Mohamed Mofreh Hamada Hamed, clinical researcher, Tanta University
Organization: Tanta University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 04-21-13
Record Dates: First submitted 2021-07-05; First posted 2021-07-12 (Actual); Last update posted 2021-07-12 (Actual); Status verified 2021-07

CONDITIONS: Tooth Extraction; Dental Implant; Extarction Socket
MeSH Terms: interventions — Blood Specimen Collection

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: statistician will be blind
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- VST with collagen plug soaked in blood (Experimental)
  Interventions: Other: VST with collagen plug soaked in blood
- VST with Allograft Demineralized bone matrix Grafton (Active Comparator)
  Interventions: Other: VST with Allograft Demineralized bone matrix Grafton
- VST with autogenous cortical chips and bovine deprotinzed particles (Active Comparator)
  Interventions: Other: VST with a particulate bone graft composed of two thirds autogenous cortical chips harvested from the surgical site and one third of bovine deprotinzed particles

INTERVENTIONS:
Other: VST with collagen plug soaked in blood — -A sub mucoperiosteal tunnel will be created, a membrane shield will be trimmed to fit the facial wall of the socket and introduced through the tunnel lying over the facial bone plate, and the facial gap will be filled with collagen plug soaked in blood
  Arms: VST with collagen plug soaked in blood
Other: VST with Allograft Demineralized bone matrix Grafton — -A sub mucoperiosteal tunnel will be created, a membrane shield will be trimmed to fit the facial wall of the socket and introduced through the tunnel lying over the facial bone plate, and the facial gap will be filled with Allograft Demineralized bone matrix Grafton
  Arms: VST with Allograft Demineralized bone matrix Grafton
Other: VST with a particulate bone graft composed of two thirds autogenous cortical chips harvested from the surgical site and one third of bovine deprotinzed particles — -A sub mucoperiosteal tunnel will be created, a membrane shield will be trimmed to fit the facial wall of the socket and introduced through the tunnel lying over the facial bone plate, and the facial gap will be filled with a particulate bone graft composed of two thirds autogenous cortical chips harvested from the surgical site and one third of bovine deprotinzed particles
  Arms: VST with autogenous cortical chips and bovine deprotinzed particles

SUMMARY:
The current research aims at evaluating the outcomes of the vestibular socket therapy in immediate implants using collagen plug, demineralized freeze-dried bone allograft, and deproteinized bovine bone minerals at both radiographic and clinical levels

ELIGIBILITY:
Inclusion Criteria:

* Patients will be included if they have one or more hopeless teeth without signs of acute infection in the maxillary anterior region.
* Remaining roots or non-restorable teeth with sufficient bone apically and palatably to allow proper implant positioning with sufficient primary stability.
* Optimal compliance as evidenced by no missed treatment appointments and a positive attitude towards oral hygiene.
* Medically free

Exclusion Criteria:

* Medically compromised patients and systemic conditions precluding implant and periodontal surgery.
* Smokers, diabetics, pregnant or lactating women.
* History of chemotherapy, radiotherapy in head and/or neck region.
* Bisphosphonate therapy

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 24 (Estimated)
Dates: Start 2021-03-16 (Actual); Primary Completion 2022-04-30 (Estimated); Study Completion 2022-07-01 (Estimated)

PRIMARY OUTCOMES:
changes in facial plate thickness | at baseline, 6 and 12 months
  Each group will be subjected to: Cone beam computed tomography (CBCT) at baseline, 6 months, and 12months to assess the thickness of the labial (facial) plate of bone and implant survival
changes in facial plate height | at baseline, 6 and 12 months
  Each group will be subjected to: Cone beam computed tomography (CBCT) at baseline, 6 months, and 12months to assess height of labial (facial) plate of bone and implant survival

SECONDARY OUTCOMES:
changes in peri-implant mucosal level | at baseline, 3rd and 6th months
  Each group will be subjected to Intraoral scanning at baseline, 6 months and 12 months. The changes in peri-implant mucosal level will be assessed by superimposition of scanning files of different intervals to monitor the changes in surface area calculated by software.

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Dentistry, Tanta University, Tanta, Egypt

REFERENCES:
- [Derived] Hamed MM, El-Tonsy MM, Elaskary A, Abdelaziz GO, Saeed SS, Elfahl BN. Effect of three different grafting materials on immediate implant placement using vestibular socket therapy in class II extraction sockets in the maxillary esthetic zone: a randomized controlled clinical trial. BMC Oral Health. 2023 Sep 1;23(1):623. doi: 10.1186/s12903-023-03345-9. PMID 37658342